CLINICAL TRIAL: NCT03977714
Title: Non-invasive Solution for Periodontal and Peri-implant Diseases
Brief Title: Non-invasive Solution for Periodontal and Peri-implant Diseases (INPERIO)
Acronym: INPERIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanoker Research S.L. (Industry)
Collaborators: Horizon 2020 - European Commission (Other); ICOA Noroeste SLP (Unknown); National Research Council, Spain (Other Government); Experior (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: INPERIO; 812065-INPERIO (Other Grant/Funding Number: EUROPEAN COMMISSION - EASME); 18/497-R_P (Other: CEIC Hospital Clínico San Carlos); 712/18/EC (Other: AEMPS)
Record Dates: First submitted 2019-05-28; First posted 2019-06-06 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Peri-Implantitis
Keywords: peri-implantitis; ceramic dental implant; non-invasive; periodontal disease; metal-free
MeSH Terms: conditions — Peri-Implantitis; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A - test implant and abutment (Experimental): Zirconia implant and G3-coated abutment (test implant and abutment). Dental sites that potentially qualify for dental implant rehabilitation will be randomly assigned to either the test group (zirconia implants) or the control group (titanium implants). Also, G3-coated and control (non-coated) abutments will be equally distributed on test and control implants, to discriminate between peri-implantitis prevention due to the G3-coating or due to the specific implant characteristics. This is a split-mouth study so that each participant can act as his or her own control and to allow between and within group comparisons.
  Interventions: Device: Zirconia implants with G3-coated abutments (test implants and abutments)
- Group B - test implant and control abutment (Experimental): Zirconia implant and control abutment (test implant, negative control abutment).
  Dental sites that potentially qualify for dental implant rehabilitation will be randomly assigned to either the test group (zirconia implants) or the control group (titanium implants). Also, G3-coated and control (non-coated) abutments will be equally distributed on test and control implants, to discriminate between peri-implantitis prevention due to the G3-coating or due to the specific implant characteristics. This is a split-mouth study so that each participant can act as his or her own control and to allow between and within group comparisons.
  Interventions: Device: Zirconia implants with control abutments (test implants, negative control abutments)
- Group C - control implant and test abutment (Experimental): Titanium implant and G3-coated abutment (control implant, test abutment). Dental sites that potentially qualify for dental implant rehabilitation will be randomly assigned to either the test group (zirconia implants) or the control group (titanium implants). Also, G3-coated and control (non-coated) abutments will be equally distributed on test and control implants, to discriminate between peri-implantitis prevention due to the G3-coating or due to the specific implant characteristics. This is a split-mouth study so that each participant can act as his or her own control and to allow between and within group comparisons.
  Interventions: Device: Titanium implants with G3-coated abutments (control implants, test abutments)
- Group D - control implant and abutment (Active Comparator): Titanium implant and control abutment (negative control implant and abutment). Dental sites that potentially qualify for dental implant rehabilitation will be randomly assigned to either the test group (zirconia implants) or the control group (titanium implants). Also, G3-coated and control (non-coated) abutments will be equally distributed on test and control implants, to discriminate between peri-implantitis prevention due to the G3-coating or due to the specific implant characteristics. This is a split-mouth study so that each participant can act as his or her own control and to allow between and within group comparisons.
  Interventions: Device: Titanium implants with control abutments (negative control implants and abutments)
- Group E - test and control implants (Experimental): Zirconia implant and titanium implant for histological and histomorphometric evaluation.
  This study will be performed in the area of the wisdom teeth (a "non useful" site that will not interfere with the rest of the study or with the patient's life), so it can only be performed in patients who no longer have these teeth. The procedure will match the procedures described for Groups A-B-C-D. Group E implants will only remain in the mouth for 2 months, after which they will be removed for further analysis. The removal of these implants, for the patient, has exactly the same implications as a normal molar extraction.
  Interventions: Device: Zirconia implants and titanium implants, for histological and histomorphometric evaluation.

INTERVENTIONS:
Device: Zirconia implants with G3-coated abutments (test implants and abutments) — Test and control interventions correspond to those usually applied in dental implantology. The "two-step protocol" will be followed. Local anesthesia will be applied. A flap will be raised to perform a progressive perforation with a gradual increase of the orifice and a profuse irrigation until the bone preparation adapts perfectly to the implant. Implants will wear a closure cap and will be covered within the gingival flap during osseointegration (eight weeks), after which they will be exposed to evaluate secondary stability and to place the abutment, for which local crestal anesthesia will be applied. To expose the closure cap, a tissue punch will generally be used. Once placed, the abutments will not be removed from the implants. All abutments will be covered with a PEEK healing cap during prosthesis fabrication. Finally, the implants will be rehabilitated with fixed prostheses according to the needs of each patient. A follow-up period of 1 year is expected.
  Arms: Group A - test implant and abutment
Device: Zirconia implants with control abutments (test implants, negative control abutments) — Test and control interventions correspond to those usually applied in dental implantology. The "two-step protocol" will be followed. Local anesthesia will be applied. A flap will be raised to perform a progressive perforation with a gradual increase of the orifice and a profuse irrigation until the bone preparation adapts perfectly to the implant. Implants will wear a closure cap and will be covered within the gingival flap during osseointegration (eight weeks), after which they will be exposed to evaluate secondary stability and to place the abutment, for which local crestal anesthesia will be applied. To expose the closure cap, a tissue punch will generally be used. Once placed, the abutments will not be removed from the implants. All abutments will be covered with a PEEK healing cap during prosthesis fabrication. Finally, the implants will be rehabilitated with fixed prostheses according to the needs of each patient. A follow-up period of 1 year is expected.
  Arms: Group B - test implant and control abutment
Device: Titanium implants with G3-coated abutments (control implants, test abutments) — Test and control interventions correspond to those usually applied in dental implantology. The "two-step protocol" will be followed. Local anesthesia will be applied. A flap will be raised to perform a progressive perforation with a gradual increase of the orifice and a profuse irrigation until the bone preparation adapts perfectly to the implant. Implants will wear a closure cap and will be covered within the gingival flap during osseointegration (eight weeks), after which they will be exposed to evaluate secondary stability and to place the abutment, for which local crestal anesthesia will be applied. To expose the closure cap, a tissue punch will generally be used. Once placed, the abutments will not be removed from the implants. All abutments will be covered with a PEEK healing cap during prosthesis fabrication. Finally, the implants will be rehabilitated with fixed prostheses according to the needs of each patient. A follow-up period of 1 year is expected.
  Arms: Group C - control implant and test abutment
Device: Titanium implants with control abutments (negative control implants and abutments) — Test and control interventions correspond to those usually applied in dental implantology. The "two-step protocol" will be followed. Local anesthesia will be applied. A flap will be raised to perform a progressive perforation with a gradual increase of the orifice and a profuse irrigation until the bone preparation adapts perfectly to the implant. Implants will wear a closure cap and will be covered within the gingival flap during osseointegration (eight weeks), after which they will be exposed to evaluate secondary stability and to place the abutment, for which local crestal anesthesia will be applied. To expose the closure cap, a tissue punch will generally be used. Once placed, the abutments will not be removed from the implants. All abutments will be covered with a PEEK healing cap during prosthesis fabrication. Finally, the implants will be rehabilitated with fixed prostheses according to the needs of each patient. A follow-up period of 1 year is expected.
  Arms: Group D - control implant and abutment
Device: Zirconia implants and titanium implants, for histological and histomorphometric evaluation. — 6 implants (3 tests and 3 controls) will be used to evaluate and compare osseointegration, via histological and histomorphometrical analysis, in the area of the wisdom teeth ("non useful" sites that will not interfere with the rest of the study or the patient's life) - it can only be performed in patients who no longer have these teeth. The procedure will match that described for Groups A-B-C-D. In this case, implants will only remain in the mouth for 2 months, after which they will be removed for analysis. The extraction will be performed with local anesthesia. A flap will be raised to expose the implant and, using a trephine bur (1 mm wider than the implant diameter), a bone cylinder containing the implant will be extracted. The resulting bone defect and regeneration process will be similar to those following a normal molar extraction. The flap will be sutured and primary curing is expected. A new implantation will not be carried out since in this area it is totally unnecessary.
  Arms: Group E - test and control implants

SUMMARY:
DESCRIPTION: The Investigational Product "A-Ce toughened TZP nanocomposite implant" is a Medical Device (MD) intended for the dental rehabilitation of edentulous sites with fixed prosthesis. The "G3®-coated NK2® abutment" is a MD intended for the prevention of peri-implant bone loss due to peri-implantitis. The MD are for dental use and will be used exclusively on subjects who have signed an informed consent form and by approved study investigators.

OBJECTIVES: (a) To evaluate the safety and performance of the "A-Ce toughened TZP nanocomposite Implant" for its intended medical application purpose in the context of successful osseointegration of zirconia-based dental implants. (b) To evaluate the safety and performance of the "G3®-coated NK2® abutment" for its intended purpose in the context of peri-implantitis prevention. (c) To obtain the regulatory CE Mark Certification status for both medical devices.

TYPE OF INVESTIGATION: Randomized double-blind (patient, appraiser) controlled study.

CENTER/COUNTRY: Instituto de Cirugía Oral Avanzada (ICOA), Madrid, Spain

GROUPS:

Group A: 30 zirconia implants with 30 G3-coated abutments (test implant and abutment) Group B: 30 test implants with 30 uncoated (control) abutments Group C: 30 Ti implants (control) with 30 test abutments Group D: 30 control implants with 30 control abutments Group E: 3 test implants and 3 control implants, for histological/histomorphometric evaluation.

COMPARATIVE DEVICE: Commercial Ti dental implant.

STATISTICAL METHODOLOGY:

H0 : INPERIO performs worse (with statistical significance) than the commercial devices.

* Test implants achieve a higher failure rate than Ti implants.
* The clinical osseointegration parameter values are worse with statistical significance for test implants than for control implants.
* Histological and histomorphometric analysis shows worse quality and quantity of osseointegration for test implants than for Ti implants.

H1: There is no statistical significance between INPERIO and the commercial solution or INPERIO performs better (with statistical significance) than the commercial Ti implants.

* Test implants achieve the same failure rate or less than Ti implants.
* The clinical osseointegration parameter values are no different or are better with statistical significance for test implants than for control implants.
* The histological and histomorphometric analysis shows a similar or better quality and quantity of osseointegration for test implants than for Ti implants.

ELIGIBILITY:
Inclusion Criteria:

* Males/females of age 18-80.
* Availability for the 18 months duration of the clinical trial.
* Subject able and willing to follow study procedures and instructions.
* Subject read, understood and signed an informed consent form.
* Participants in need of dental implant treatment and that meet one of the following criteria:

  * Moderate to advanced periodontitis.
  * History of dental loss attributed to periodontitis.
  * Risk factors associated with periodontitis (tobacco consumption, poor oral hygiene, diabetes patients outside of the ideal range control (HbA1c <7)).
* Good general health at time of inclusion.
* Subjects willing to disclose information on medication.

Exclusion Criteria:

* Female patients who report being pregnant or lactating, or who are of childbearing potential and are not using hormonal, barrier methods of birth control or abstinence.
* Subject chronically treated (≥ two weeks) with any medication known to affect inflammation or periodontal status six months prior to enrollment or during the study.
* Subject necessitating antibiotic for 1 month during the study.
* Gross oral pathology.
* Participation in any other clinical study or test panel within one month prior to entry into the study.
* History of neoplastic disease requiring the use of chemotherapy.
* Patients with history of renal failure or chronic renal diseases.
* Patients affected by chronic liver diseases.
* Patients with severe or uncontrolled metabolic bone disorders.
* Conditions or circumstances, in the opinion of the investigator, which could represent a general contra-indication for undergoing surgery, or could prevent study completion or interfere with the analysis of the results, such as a history of non-compliance or unreliability.
* History of local radiation therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Implant performance verification: implant survival rate. Change will be assessed. | Day 1 (abutment connection), 3 months, 6 months, 1 year.
  Number of functional implants vs. number of implants inserted.
Implant performance verification: osseointegration (in vivo). Change will be assessed. | Day 1 (abutment connection), 3 months, 6 months, 1 year.
  Osseointegration quality: implant stability will be assessed via metal instrument tapping - the transmitted sound will indicate good/bad osseointegration.
Implant performance verification: osseointegration (in vivo). Change will be assessed. | Day 1 (abutment connection), 3 months, 6 months, 1 year.
  Osseointegration quantity: distance from the implant platform to the first bone contact (assessed via probing).
Implant performance verification: osseointegration (in vivo). Change will be assessed. | Day 1 (abutment connection), 3 months, 6 months, 1 year.
  Osseointegration quantity: bone to implant contact (BIC) (assessed via standard parallel periapical radiographs).
Implant performance verification: osseointegration (in vivo). Change will be assessed. | Day 1 (abutment connection), 3 months, 6 months, 1 year.
  Osseointegration quantity: bone density/quality (assessed via standard parallel periapical radiographs).
Implant performance verification: osseointegration (ex vivo). | 2 months after implantation.
  Please refer to Arms and Interventions, Experimental: Group E. For ethical reasons, this sample size is limited to six (6) implants, 3 test and 3 controls. Trephined blocks containing the explanted implants will be stored in a 5% formaldehyde solution (pH 7). They will be immersed in a 4% formaldehyde and 1% calcium solution and processed for ground sectioning following the Donath & Breuner methods. Each implant block will be individualized, embedded in methyl-methacrylate and stained with combined Harris Haematoxyline and Wheatley. The analysis will be performed using a transmitted light microscope equipped with a digital camera. Results will be inferred to clinical osseointegration data, which is the way to assess osseointegration in everyday chairside practice.
G3-coated abutment performance in peri-implantitis prevention. Change will be assessed. | Day 1 (abutment connection), 3 months, 6 months, 1 year.
  Assessment of peri-implant inflammation sign: bleeding on probing (BOP).
G3-coated abutment performance in peri-implantitis prevention. Change will be assessed. | Day 1 (abutment connection), 3 months, 6 months, 1 year.
  Assessment of gingival alteration sign: gingival clinical attachment level (CAL). Peri-implantitis is defined as bone loss around implants, so crestal bone loss will be assessed using the gold standard parallel X-Ray technique to evaluate any changes in bone to implant contact (BIC) at both mesial and distal aspects of all implants.
G3-coated abutment performance in peri-implantitis prevention. Change will be assessed. | Day 1 (abutment connection), 3 months, 6 months, 1 year.
  Assessment of crestal bone loss. Peri-implantitis is defined as bone loss around implants, so crestal bone loss will be assessed using the gold standard parallel X-Ray technique to evaluate any changes in bone to implant contact (BIC) at both mesial and distal aspects of all implants.

SECONDARY OUTCOMES:
Prosthetic complications. Change will be assessed. | Day 1 (abutment connection), 3 months, 6 months, 1 year.
  Assessment of parameters that may act as predisposing factors for prosthetic complications (checklist: smoker; drinking habits, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto López Píriz, MD, DDS, PhD, Principal Investigator — ICOA Noroeste SLP
Locations (1):
- ICOA Noroeste SLP, Las Rozas de Madrid, Madrid, Spain